CLINICAL TRIAL: NCT06307366
Title: Perceptions and Experiences of (Future) Parents With Mental Illness and Family Members of People With Mental Illness About Risk for Mental Illness in (Future) Children, Potential Resilience Factors, and Needs for Care and Research
Brief Title: Perceptions and Experiences of (Family Members of) People With Mental Illness About the Chance for Mental Illness in (Future) Children, and Needs for Care and Research
Acronym: PANDAcc
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Lisanne van Houtum, Postdoctoral researcher designated by Prinicipal Investigator, Erasmus Medical Center
Other Study IDs: ErasmusMC10365
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Mental Illness
Keywords: mental illness; risk; resilience; offspring; qualitative research; mood-psychosis spectrum
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- (Future) parents with (a partner with) mental illness in the mood-psychosis spectrum: The following participants will be included: (Future) parents with (a partner with) mental illness in the mood-psychosis spectrum (psychotic disorder, bipolar disorder, severe depression); ≥ 18 years old.
  If including (future) parents with mental illness and their partners will turn out to be difficult given our timeframe, we will mitigate this by additionally including family members of people with mental illness, e.g. siblings or grandparents.
  Interventions: Other: No intervention will be used

INTERVENTIONS:
Other: No intervention will be used — This is a qualitative study, no intervention will be used

SUMMARY:
Despite consistent evidence that mental illness runs in families, intergenerational transmission of risk of mental illness is rarely considered in clinical practice. Neither preventive programs for children of parents with mental illness are usually implemented in care, nor supportive programs for parenting. Furthermore, parents with mental illness are not always aware of how their disorder may impact the well-being of their children. To date, the needs for counseling, care and research in parents with mental illness and family members of people with mental illness are unclear. Therefore, this prospective qualitative interview study aims to gain insights into the perceptions and experiences of (future) parents with mental illness, partners and family members of people with mental illness about risk for and resilience against mental illness in (future) children, as well as their needs for counseling, care and research.

ELIGIBILITY:
Inclusion Criteria:

* Having (a partner or relative with) a diagnosis of a mental illness in the mood-psychosis spectrum, i.e., psychotic disorder, bipolar disorder, or severe depression
* At least 18 years old

Exclusion Criteria:

* Insufficient proficiency of the Dutch language
* No demonstration of adequate understanding of the purpose, procedures, risks, benefits, emergency contacts, and payment issues (in accordance with criteria to assess capacities to consent from Appelbaum & Grisso, 1988).
* Unable to give consent to all aspects of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The following participants will be included: (Future) parents with (a partner with) mental illness in the mood-psychosis spectrum (psychotic disorder, bipolar disorder, severe depression); ≥ 18 years old.
  If including (future) parents with mental illness and their partners will turn out to be difficult given our timeframe, we will mitigate this by additionally including family members of people with mental illness, e.g. siblings or grandparents.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Themes around the topics (related to perceptions and experiences) explored. | 1 hour
  We developed an interview guide around the main themes (i) risk and resilience; (ii) information needs for care and counselling; and (iii) (biological) research to ensure key aspects relating to perceptions, experiences, and needs of participants around the chance risk for mental illness in (future) children will be covered during the interviews. It additionally allows the interviewer to ask follow-up questions on interesting perspectives put forth by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Hilmar H. Bijma, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Only processed, group-level data (i.e., themes, subthemes) can be shared, given that interviews can be traced back to individual participants. The PI will verify the authenticity of the requesting researcher and will check whether their intentions are in line with the informed consent and whether the intended methodology is suitable and will approve the request before providing access to the data.
  A Data Transfer Agreement will be signed, and the Technology Transfer Office will be involved to ensure the appropriate agreements are made.